CLINICAL TRIAL: NCT01380951
Title: Clinical Study of Telbivudine on Liver Cirrhosis in Patients With Chronic Hepatitis B
Brief Title: Safety and Efficacy of Telbivudine on Liver Cirrhosis in Patients With Chronic Hepatitis B (CHB)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Fifth People's Hospital of Suzhou (Other)
Responsible Party: Chuanwu Zhu, the Fifth People's Hospital of Suzhou
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: szwy20110610
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Liver Cirrhosis; Chronic Hepatitis B
Keywords: liver cirrhosis; chronic hepatitis B; antiviral therapy; telbivudine
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis B, Chronic | interventions — Telbivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- telbivudine (Experimental)
  Interventions: Drug: telbivudine

INTERVENTIONS:
Drug: telbivudine — telbivudine 600mg/d 96 weeks
  Other Names: Sebivo

SUMMARY:
Antiviral treatment on Chronic Hepatitis B (CHB) patients with liver cirrhosis is compulsory and effective. Telbivudine, which is superior to lamivudine in the treatment of CHB,is considered to be appropriate for the antiviral treatment on CHB patients with liver cirrhosis.

DETAILED DESCRIPTION:
Antiviral therapy on CHB patients with liver cirrhosis is compulsory and effective. Diseases development can be prevented or delayed if the virus is depressed successfully. Lamivudine is often used and usually has good efficacy. However, lamivudine resistance and virus mutation happens a lot. Telbivudine, which is superior to lamivudine in the treatment of CHB,is considered to be appropriate for the antiviral treatment on CHB patients with liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* liver cirrhosis with CHB
* without history of antiviral therapy or discontinued antiviral therapy for more than 6 months
* for patients with compensated liver cirrhosis: HBV DNA≥4log copies/ml if HBeAg positive,HBV DNA≥3log copies/ml if HBeAg negative
* for patients with uncompensated liver cirrhosis:HBV DNA positive

Exclusion Criteria:

* coinfection with HCV,HDV and HIV
* AFP≥100mg/L or HCC diagnosed by iconography
* with severe cardiovascular, respiratory and endocrinology diseases or autoimmune diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Serum HBV DNA | 48 weeks
  serum HBV DNA negativity and decline from baseline at week 48

SECONDARY OUTCOMES:
Serum HBeAg | 48 weeks
  rate of HBeAg seroconversion and HBeAg loss
Child-pugh score | 48 weeks
  the average decline of Child-pugh score at week 48 from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Chuanwu Zhu, Doctor, Principal Investigator — The Fifth People's Hospital of Suzhou
Locations (1):
- the Fifth People's Hospital of Suzhou, Suzhou, Jiangsu, China